CLINICAL TRIAL: NCT07036861
Title: A Comparative Bioavailability of Reformulated Ibuprofen 2% and 4% Oral Suspensions (Berlin Chemie AG) and Reference Ibuprofen (Nurofen®) 200 mg/5 ml Oral Suspension in Healthy Male and Female Adult Subjects Under Fasting Conditions: an Open-label, Randomized, Single-dose, Three-period, Three-treatment, Three-sequence Crossover Study
Brief Title: A Comparative Bioavailability Study of Reformulated Ibuprofen 2% and 4% Oral Suspensions (Berlin Chemie AG) and Versus Ibuprofen (Nurofen®) 200 mg/5 ml Oral Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BCLT/22/IBU-BE/001; 2023-503703-28 (EudraCT Number)
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy Male and Female Subjects
Keywords: Ibuprofen oral suspension; Nurofen oral suspension; Bioequivalence study

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, single-dose, three-period, three treatment, three sequence crossover bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen 2% oral suspension (T1), reformulated (Experimental): 400 mg to be taken with a graded syringe
  Interventions: Drug: Ibuprofen 2%
- Ibuprofen 4% oral suspension (T2), reformulated (Experimental): 400 mg to be taken with a graded syringe
  Interventions: Drug: Ibuprofen 4%
- Nurofen dla dzieci Forte pomarańczowy 40 mg/mL, oral suspension, Reckitt-Benckiser (Poland) S.A. (Active Comparator): 400 mg to be taken with a graded syringe
  Interventions: Drug: Ibuprofen 4%

INTERVENTIONS:
Drug: Ibuprofen 2% — Reformulated Ibuprofen 2% oral suspension (Berlin-Chemie AG)
  Arms: Ibuprofen 2% oral suspension (T1), reformulated
Drug: Ibuprofen 4% — Reformulated Ibuprofen 4% oral suspension (Berlin-Chemie AG)
  Arms: Ibuprofen 4% oral suspension (T2), reformulated
Drug: Ibuprofen 4% — Nurofen dla dzieci Forte pomarańczowy 40 mg/mL, oral suspension (Polish brand name)
  Arms: Nurofen dla dzieci Forte pomarańczowy 40 mg/mL, oral suspension, Reckitt-Benckiser (Poland) S.A.

SUMMARY:
Purpose of the study is to compare three different formulations of Ibuprofen oral suspension (liquid taken by mouth) to see if there are any differences in how much of the active substance and how quickly it was taken up by by the body, broken down, and how quickly it was removed from the body.

DETAILED DESCRIPTION:
In this Phase 1 study, two test medications (reformulated Ibuprofen 2% oral suspension and Ibuprofen 4% oral suspension) were compared with the reference medication (Ibuprofen 4% oral suspension marketed under the trade name Nurofen dla dzieci Forte pomarańczowy 40 mg/mL, oral suspension) in terms of bioequovalence of the tested formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the informed consent form (ICF) and giving signed informed consent which includes compliance with the requirements and restrictions as listed in the ICF and the study protocol.
2. Healthy male and female subjects aged 18 to 45 years inclusive at the time of ICF signature.
3. Healthy as determined by an Investigator based on the results of the standard clinical, laboratory and instrumental methods of examination.
4. Body weight ≥ 50 kg and Body Mass Index (BMI) between ≥ 18.5 and ≤ 30 kg/m2.
5. Non-smokers (for at least 3 months before screening) verified by a cotinine test at screening.
6. A negative urine pregnancy test (rapid test) within 24 hours before the first IMP dose for female subjects of childbearing potential.

   Postmenopausal (no menses for at least 1 year) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) female subjects are exempted from this requirement.
7. Subjects with preserved reproductive potential agree to use, with their partner, adequate contraception throughout the study and for 15 days thereafter (contraceptive methods with reliability greater than 90%: cervical caps with spermicide, diaphragms with spermicide, condoms with intravaginal spermicide, oral, injectable, transdermal or implanted hormonal contraceptives, vaginal contraceptive ring, non-hormonal intrauterine devices), or true sexual abstinence.

Exclusion Criteria:

1. History or presence of allergies.
2. Known hypersensitivity or intolerance to ibuprofen or other non-steroidal anti-inflammatory drugs (NSAIDs), fructose and/or any excipient of the IMP.
3. History of bronchospasm, asthma, rhinitis, angioedema or urticaria associated with the intake of acetylsalicylic acid or other NSAIDs.
4. History or presence of significant cardiovascular (including congestive heart failure (NYHA IV), arterial hypertension, established ischemic heart disease, peripheral arterial disease, and/or cerebrovascular disease), pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, infectious, dermatologic, neurologic, or psychiatric disease.
5. History of recurrent peptic ulcer or gastrointestinal bleeding (>2 distinct episodes of proven ulceration or bleeding) or history of gastrointestinal bleeding or perforation related to previous NSAID therapy.
6. Cerebrovascular or other active bleeding.
7. Acute infectious diseases of any organ system (including e.g., influenza, COVID-19, acute respiratory viral infections) less than 4 weeks before the first IMP dose.
8. History or presence of any other clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
9. History of major abdominal surgery or minor abdominal surgery within 3 months before the first IMP dose.
10. Clinically significant deviations from the normal parameters (see study protocol Appendix 2 for guidance) in clinical blood count analysis, biochemical blood analysis, urinalysis.
11. Systolic blood pressure measured in a supine position < 100 mmHg or > 130 mmHg and/or diastolic blood pressure < 60 mmHg or > 89 mmHg.
12. Heart rate < 60 or > 100 beats per minute.
13. Female subjects who were attempting to conceive, pregnant or lactating.
14. Positive test results for HIV or hepatitis B (HBsAg, anti-HBc) or hepatitis C (anti-HCV) or syphilis at screening.
15. Positive screen for drugs of abuse or alcohol at screening.
16. Positive test result for cotinine in urine at screening.
17. Known or suspected drug or alcohol abuse as judged by the Investigator.
18. Alcohol consumption more than 10 units of alcohol a week (1 unit = 200 mL of dry wine or 50 mL of strong alcoholic drinks or 500 mL of beer) within 6 months before the first IMP dose.
19. Intake of methylxanthine containing substances (e.g., coffee, tea, chocolate, cocoa, energy drinks, cola) as well as citrus fruits and cranberry (including juices, fruit drinks, etc.) within the last 24 h before the first IMP dose.
20. Intake of medications that had a significant effect on circulatory dynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, NSAIDs, angiotensin-converting enzyme inhibitors, angiotensin II receptor antagonists, diuretics, etc.) within the 2 months before the first IMP dose.
21. Use of any prescribed or nonprescribed medication, herbal remedies, vitamins and minerals within the 2 weeks before the first IMP dose or longer (at least 5 elimination half-lives) if the medication has a long half-life.
22. Mental, physical and other reasons that did not allow the subjects according to Investigator's opinion to assess their behavior adequately, to follow correctly the requirements of the clinical study protocol and to assess the expected risks and possible discomfort.
23. Dehydration (e.g. due to diarrhea, vomiting, or other causes) within the last 48 h before the first IMP dose.
24. Subjects who had been on a special diet (for whatever reason, e.g., vegetarians or hypocaloric diet [< 1000 kcal/day]) within the 28 days before the first IMP dose.
25. Plasma donation within 1 month of screening or blood donation/blood loss >500 mL within the 3 months before screening.
26. Unwillingness or inability to follow the procedures and restrictions outlined in the protocol and the ICF.
27. Participation in another clinical study within the 3 months before the first IMP dose in this study.
28. Female subjects with childbearing potential, having unprotected sexual intercourse with any unsterilized male partner (i.e., a man who is not sterilized by vasectomy for at least 6 months) within the 30 days before the first IMP dose.
29. Any reason in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Cmax | 24 hours
  Maximum plasma concentration
AUC0-t | 24 hours
  Area under the curve
tmax | 24 hours
  Time to maximum plasma concentration

SECONDARY OUTCOMES:
AUC0-inf | 24 hours
  Area under the curve to infinity
Residual area | 24 hours
λz | 24 hours
  elimination constant
t1/2 | 24 hours
  Half-life

OTHER OUTCOMES:
Safety evaluation | 45 days
  Incidence and type of Adverse Events (AEs)
Safety evaluation | 45 days
  Proportion of subjects with treatment-related adverse events
Safety evaluation | 45 days
  Proportion of subjects experiencing Serious Adverse Events (SAEs)
Safety evaluation | 45 days
  Proportion of subjects with treatment-related SAEs
Safety evaluation | 45 days
  Proportion of subjects discontinued from the study due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Greta Burneikaitė, MD, PhD, Principal Investigator — Vilnius University Hospital Santaros Klinikos
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No
No publication in an ICMJE journal is planned

REFERENCES:
- See also: Related Info — https://www.menarini.com/en-us/innovation-research/clinical-trials/clinical-trials-database